CLINICAL TRIAL: NCT03655340
Title: A 24-month Prospective, Non-interventional, Multicentre Study to Evaluate the Real-world Effectiveness and Usage of Alprolix in Patients With Haemophilia B in France
Brief Title: A Study to Evaluate the Real-world Effectiveness and Usage of Alprolix in Patients With Haemophilia B in France
Acronym: B-SURE
Status: Completed | Type: Observational
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Other Study IDs: Sobi.Alprolix-001
Record Dates: First submitted 2018-08-30; First posted 2018-08-31 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Haemophilia B
Keywords: Blood Coagulation Disorder; Hematologic Diseases; Coagulation Protein Disorder; Hemorrhagic Disorder; Genetic Diseases, Inborn
MeSH Terms: conditions — Hemophilia B; Blood Coagulation Disorders; Hematologic Diseases; Coagulation Protein Disorders; Hemorrhagic Disorders; Genetic Diseases, Inborn | interventions — factor IX Fc fusion protein

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prophylactic patients: Alprolix will be prescribed according to local practice and administered by patients with haemophilia B for prophylactic treatment
  Interventions: Drug: Alprolix
- On demand patients: Alprolix will be prescribed according to local practice and administered by patients with haemophilia B for on-demand treatment
  Interventions: Drug: Alprolix

INTERVENTIONS:
Drug: Alprolix — Extended half-life factor IX product
  Other Names: Eftrenonacog alfa, rFIXFc

SUMMARY:
Alprolix (rFIXFc) is a recombinant extended half-life coagulation factor product. The purpose of this non-interventional study is to describe the real-world usage and effectiveness of Alprolix in the on-demand and prophylactic treatment of haemophilia B.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of haemophilia B and been treated previously with factor IX Product
* Have started Alprolix treatment prior to enrolment visit, or at enrolment prescribed treatment with Alprolix, regardless of participation in the study
* Signed and dated informed consent provided by the patient, or the patient's legally acceptable representative for patients under the legal age, before any study-related activities are undertaken. Assent should be obtained from paediatric patients according to local regulations

Exclusion Criteria:

* Participation in an investigational medicinal product trial at enrolment visit

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All eligible patients who present for a routine Clinical visit will be asked to participate in the study by the treating physician at participating haemophilia treatment centres in France.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
Annualised bleeding rate (ABR) (prophylactic treatment) | 24 months
  Assessed by diary
Annualised injection frequency (prophylactic treatment) | 24 months
  Assessed by diary
Annualised factor consumption (International Unit [IU]) (prophylactic treatment) | 24 months
  Assessed by diary
Amount of factor Product used to treat a bleed (on-demand treatment) | 24 months
  Assessed by diary
Number of injections to treat a bleed (on-demand treatment) | 24 months
  Assessed by diary

CONTACTS AND LOCATIONS:
Overall Officials: Elena Santagostino, MD, Study Director — Swedish Orphan Biovitrum
Locations (18):
- France (18):
  - Swedish Orphan Biovitrum Research Site (CHU de Bordeaux), Bordeaux
  - Swedish Orphan Biovitrum Research Site, Brest
  - Swedish Orphan Biovitrum Research Site, Caen
  - Swedish Orphan Biovitrum Research Site, Chambéry
  - Swedish Orphan Biovitrum Research Site, Clermont-Ferrand
  - Swedish Orphan Biovitrum Research Site, Dijon
  - Swedish Orphan Biovitrum Research Site, La Réunion
  - Swedish Orphan Biovitrum Research Site, Lille
  - Swedish Orphan Biovitrum Research Site, Marseille
  - Swedish Orphan Biovitrum Research Site, Montpellier
  - Swedish Orphan Biovitrum Research Site, Nantes
  - Swedish Orphan Biovitrum Research Site, Nîmes
  - Swedish Orphan Biovitrum research site, Paris
  - Swedish Orphan Biovitrum research site, Poitiers
  - Swedish Orphan Biovitrum research site, Rennes
  - Swedish Orphan Biovitrum Research Site, Rouen
  - Swedish Orphan Biovitrum research site, Strasbourg
  - Swedish Orphan Biovitrum Research Site, Toulouse

REFERENCES:
- [Derived] Chambost H, Repesse Y, Genre-Volot F, Desprez D, Castet SM, Vanderbecken S, Zidi M, Gandossi C, Nuesch E, Palmborg H, Santagostino E; B-SURE Study Group. Real-world usage and effectiveness of recombinant factor IX Fc in haemophilia B from the B-SURE study in France. Ther Adv Hematol. 2025 Jan 26;16:20406207241311535. doi: 10.1177/20406207241311535. eCollection 2025. PMID 39872008